CLINICAL TRIAL: NCT00408564
Title: Phase II Study of Neoadjuvant Gemcitabine/Oxaliplatin and Cetuximab Followed by Surgery or Concurrent External Beam Radiation With Capecitabine for Patients With Locally Advanced Unresectable Nonmetastatic Pancreatic Cancer
Brief Title: Cetuximab, Gemcitabine, and Oxaliplatin Followed By Surgery or External-Beam Radiation Therapy and Capecitabine in Treating Patients With Locally Advanced, Nonmetastatic Pancreatic Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000518313; MUSC-100918; BMS-MUSC-100918; SANOFI-MUSC-100918
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-05

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage II pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Capecitabine; Oxaliplatin; Radiotherapy; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine,Oxaliplatin and Cetuximab (Experimental): Gemcitabine will be given on day 1 of every 2 week cycle. Oxaliplatin will be given day 2 of every 2 week cycle. Cetuximab will be given every week for 12 weeks.
  After chemotherapy, patient will be assessed for resectability. Patients will have either surgery or daily radiation and capceitabine Monday-Friday for a total of 5 and a half weeks.
  Interventions: Biological: cetuximab; Drug: capecitabine; Drug: oxaliplatin; Procedure: conventional surgery; Radiation: radiation therapy; Drug: Gemcitabine

INTERVENTIONS:
Biological: cetuximab
Drug: capecitabine
Drug: oxaliplatin
Procedure: conventional surgery
Radiation: radiation therapy
Drug: Gemcitabine

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as gemcitabine, oxaliplatin, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sometimes when chemotherapy is given, it does not stop the growth of tumor cells. The tumor is said to be resistant to chemotherapy. Giving cetuximab together with chemotherapy may reduce drug resistance and allow the tumor cells to be killed. Giving cetuximab and chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Radiation therapy uses high-energy x-rays to kill tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with oxaliplatin and gemcitabine followed by surgery or external-beam radiation therapy and capecitabine works in treating patients with locally advanced, nonmetastatic pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the progression-free survival rate in patients with unresectable, locally advanced, nonmetastatic adenocarcinoma of the pancreas treated with neoadjuvant therapy comprising cetuximab, gemcitabine hydrochloride, and oxaliplatin followed by either surgery or chemoradiotherapy comprising external-beam radiotherapy and capecitabine.

Secondary

* Determine the toxicity and tolerability of this regimen in these patients.
* Determine overall survival and progression-free survival.
* Determine the response rate in these patients.
* Determine the response duration (defined as the time from first observation response to the time of progressive disease) in patients who achieve at least a partial response to treatment.
* Determine the biomarker response of CA19-9.

OUTLINE: This is an open-label study.

* Neoadjuvant therapy: Patients receive cetuximab IV over 1-2 hours on days 1 and 8, gemcitabine hydrochloride IV over 100 minutes on day 1, and oxaliplatin IV over 2 hours on day 2. Treatment repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are evaluated after completion of neoadjuvant therapy. Patients with metastatic disease are taken off study. Beginning within 4 weeks after completion of neoadjuvant therapy, patients with resectable disease proceed to surgical resection or chemoradiotherapy (by choice); patients with unresectable disease proceed to chemoradiotherapy.

* Surgery: Patients undergo surgical resection with the Whipple procedure.
* Chemoradiotherapy: Patients receive oral capecitabine twice daily 5 days a week (on days 1-5) and undergo external-beam radiotherapy once daily 5 days a week for 5½ weeks.

After completion of study treatment, patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or radiologically confirmed pancreatic cancer, meeting both of the following criteria:

  * Locally advanced, nonmetastatic disease
  * Surgically unresectable disease
* Measurable disease, defined as unidimensionally measurable by physical exam or imaging study

  * The following are considered nonmeasurable disease:

    * Bone-only disease
    * Pleural or peritoneal effusions
    * CNS lesions
    * Irradiated lesions in the absence of progression after radiotherapy
* No history or evidence of CNS disease
* No metastatic disease to distant organs (e.g., liver, lung, brain, or bone)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 2.0 mg/dL
* Creatinine ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 90 days after completion of study therapy
* No acute hepatitis
* No known HIV positivity
* No active or uncontrolled infection
* No significant history of uncontrolled cardiac disease, including, but not limited to, any of the following:

  * Uncontrolled hypertension
  * Unstable angina
  * Myocardial infarction within the past 6 months
  * Uncontrolled congestive heart failure
  * Cardiomyopathy with decreased ejection fraction
* No prior severe infusion reaction to a monoclonal antibody
* No active second malignancy other than nonmelanoma skin cancer
* No history of deep vein thrombosis
* No history of bleeding diathesis or coagulopathy
* No other severe concurrent disease, mental incapacitation, or psychiatric illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

* No prior therapy for pancreatic cancer
* No prior therapy specifically targeting the epidermal growth factor-receptor pathway
* No major surgical procedure or open biopsy within the past 28 days
* No prior radiotherapy or chemotherapy
* No prior or concurrent full-dose anticoagulants or thrombolytics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S. Kraft, MD, Principal Investigator — Medical University of South Carolina; Gustavo Leone, Study Chair — Medical University of South Carolina, Hollings Cancer Center
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine,Oxaliplatin and Cetuximab: Gemcitabine will be given on day 1 of every 2 week cycle. Oxaliplatin will be given day 2 of every 2 week cycle. Cetuximab will be given every week for 12 weeks.
  After chemotherapy, patient will be assessed for resectability. Patients will have either surgery or daily radiation and capceitabine Monday-Friday for a total of 5 and a half weeks.
  cetuximab
  capecitabine
  oxaliplatin
  conventional surgery
  neoadjuvant therapy
  radiation therapy
  Gemcitabine
Period: Overall Study
Arm/Group | Gemcitabine,Oxaliplatin and Cetuximab
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine,Oxaliplatin and Cetuximab
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months
Time Frame: up to 46 weeks after the start of study treatment
Population: only includes patients who completed at least 2 cycles of induction chemotherapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine,Oxaliplatin and Cetuximab
Number analyzed (Participants) | 38
percentage of participants | 82 [70 to 95]

2. Secondary Outcome: Number of Participants With Grade 3-4 Adverse Events Reported
Time Frame: from start of study treatment until end of study visit, about 30 weeks
Measure: Number; unit: participants
Arm/Group | Gemcitabine,Oxaliplatin and Cetuximab
Number analyzed (Participants) | 39
participants | 9

3. Secondary Outcome: Overall Survival
Time Frame: up to 46 weeks after the start of study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine,Oxaliplatin and Cetuximab
Number analyzed (Participants) | 38
percentage of participants | 49 [36 to 68]

4. Secondary Outcome: Response Rate
Description: defined as the total number of subjects whose best response is PR or CR.
Time Frame: up to 46 weeks after the start of study treatment
Population: only includes patients who completed at least 2 cycles of induction chemotherapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine,Oxaliplatin and Cetuximab
Number analyzed (Participants) | 38
Participants | 5

5. Secondary Outcome: Response Duration in Patients With at Least Partial Response to Treatment
Time Frame: up to 46 weeks after the start of study treatment
Population: data for this endpoint was not collected.
Arm/Group | Gemcitabine,Oxaliplatin and Cetuximab
Number analyzed (Participants) | 0

6. Secondary Outcome: Determine the Biomarker Response of CA 19-9 to Therapy
Time Frame: from start up treatment to one year after end of treatment, up to 81 weeks
Population: data for this endpoint was not collected.
Arm/Group | Gemcitabine,Oxaliplatin and Cetuximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events will be assessed from the start of study therapy until the end of therapy visit (up to 13 weeks).
Description: "Other adverse event" information is not available for reporting.
Arm/Group | Gemcitabine,Oxaliplatin and Cetuximab
Serious Adverse Events (participants affected / at risk) | 13/39
Other Adverse Events (participants affected / at risk) | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine,Oxaliplatin and Cetuximab (N=39)
vomiting (Gastrointestinal disorders) | 6
metabolic acidosis (Investigations) | 2
respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
fractured right arm (Musculoskeletal and connective tissue disorders) | 1
abdominal pain (Gastrointestinal disorders) | 2
urinary tract infection (Renal and urinary disorders) | 1
weakness (Musculoskeletal and connective tissue disorders) | 2
bradycardia (Cardiac disorders) | 1
dehydration (Gastrointestinal disorders) | 2
billiary obstruction (Renal and urinary disorders) | 2
fever (General disorders) | 1
fall (General disorders) | 2
anorexia (Gastrointestinal disorders) | 1
edema (General disorders) | 1
jaundice (Hepatobiliary disorders) | 1
altered mental status (Psychiatric disorders) | 1
pain (Musculoskeletal and connective tissue disorders) | 1
nausea (Gastrointestinal disorders) | 6
weight loss (General disorders) | 1
diarrhea (Gastrointestinal disorders) | 2
hypokalemia (Metabolism and nutrition disorders) | 2
fecal impaction (Gastrointestinal disorders) | 1
allergic reaction (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No